CLINICAL TRIAL: NCT01092221
Title: Allopurinol for Mania: A Randomized Trial Administering Allopurinol vs. Placebo as add-on to Mood Stabilizers and/or Antipsychotics in Patients in a Bipolar Manic Episode.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHEBA-10-7724-MW-CTIL
Record Dates: First submitted 2010-03-17; First posted 2010-03-24 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Mania
Keywords: mania, allopurinol, add-on treatment
MeSH Terms: conditions — Mania | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allopurinol (Experimental)
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allopurinol — Allopurinol 1 capsule 300 mg, BID
  Other Names: Alloril, Zylol, Zyloric
  Arms: Allopurinol
Drug: Placebo — Placebo 1 capsule, 300 mg, BID
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the efficacy of allopurinol, compared to placebo, as add-on to mood stabilizers and/or antipsychotic in the treatment of patients with bipolar disorder, in a manic episode.

DETAILED DESCRIPTION:
An emerging body of evidence supports a role for dysfunctional purinergic related neurotransmission in mood disorders [1, 2]. Adenosine agonists have been shown to have properties similar to those of dopamine antagonists and there is a well characterized antagonistic interaction between adenosine and dopamine receptors in the ventral striatum. Increased adenosynergic transmission has been demonstrated to reduce the affinity of dopamine agonists for dopamine receptors. It has been theorized that adenosine may exert some of its antipsychotic effects through modulation of glutamatergic transmission.

Two double-blind, randomized, add-on, placebo-controlled trials comparing allopurinol and placebo in acute mania have showed statistically significant greater improvements in YMRS scores in the allopurinol vs. placebo groups. These empiric data, together with the theoretical and basic science background cited, provide the impetus for this proposed study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-65 years of age, inclusive
2. Only females who are abstinent or practicing an established method of birth control (oral contraceptive tablets, hormonal implant device, hormone patch, injectable contraceptive, intrauterine device [IUD]) can be included in the trial.
3. Willing and able to provide informed consent, after the nature of the study has been fully explained
4. Current DSM-IV-TR diagnosis of bipolar I disorder with the current episode manic (296.4x) or mixed (296.6x), as confirmed by the Modified Structured Clinical Interview for DSM-IV (SCID). In order to ensure that this is an acute manic episode, we will verify that the current manic episode was preceded by a period of euthymia or depression. If inpatients, subjects will be included only up to 14 days after admission. Subjects with psychotic features will be included in the study.
5. YMRS> 17
6. Patients receiving one or multiple mood stabilizers, and/or one or more anti-psychotics.
7. Inpatients or outpatients.

Exclusion Criteria:

1. Unwilling or unable, in the opinion of the Investigator, to comply with study instructions
2. Pregnant or breast-feeding
3. Unstable medical disease (malignancy, poorly controlled diabetes, active ischemic cardiac disease, or cardiomyopathy, serious pulmonary disease, kidney disease, impaired liver functioning).
4. Currently taking any of the following medications: warfarin, amoxicilline, ampicilline, theophylline, or mycophenolate mofetil.
5. Likely allergy or sensitivity to Allopurinol
6. At significant risk of committing suicide, or in the opinion of the Investigator, currently is at imminent risk of suicide or harming others.
7. Suffers from a significant Substance Dependence disorder based on DSM-IV criteria within the 3 months prior to Screening, or is deemed by the Investigator to have a high risk of substance use during the study. Patients with a history of recreational use of cannabinoids or alcohol, and/or patients who smoke cigarettes can be included.
8. Concurrent delirium, mental retardation, drug-induced psychosis, or history of brain trauma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
1) Change from baseline to day 42 in the YMRS | from baseline to day 42
2) Change from baseline to day 42 in the CGI-BP scale. | from baseline to day 42

SECONDARY OUTCOMES:
1) Change from baseline to day 14 in the YMRS | from baseline to day 14
2) Change from baseline to day 14 in the CGI-BP scale. | from baseline to day 14
3) Change in the PANSS activation subscale score (total score of 6 PANSS items: Hostility, poor impulse control, excitement, uncooperativeness, poor rapport, and tension) from baseline to final assessment (Day 42). | from baseline to day 42
4) Rates of discontinuation in the allopurinol group compared to the placebo group | during the study period (42 days)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Weiser, Principal Investigator — Sheba Medical Center
Locations (24):
- Israel (3):
  - Beer-Yaakov Mental Health Center, Beer-Yaakov
  - Sheba Medical Center, Ramat Gan
  - Lev Hasharon Mental Health Center, Tsur Moshe
- Romania (21):
  - Spitalul de Psihiatrie, si Neurologie, Brasov, Brasov, Brașov County
  - Spitalul Clinic de Psihiatrie "Prof.Al. Obregia" Sectia 12, Bucharest, Bucharest
  - Spitalul Clinic de Psihiatrie "Prof.Al. Obregia" Sectia 1, Bucharest, Bucharest
  - Spitalul Clinic de Psihiatrie "Prof.Al. Obregia" Sectia 3, Bucharest, Bucharest
  - Spitalul Clinic Judetean, de Urgenta,, Cluj-Napoca, Cluj-Napoca
  - Sp. Judetean, Focşani, Focsani
  - Sp de Psihiatrie Galati, Galati, Galați County
  - Spitalul Clinic de Psihiatrie, "Socola",, Iași, Iaşi
  - Spitalul Clinic de Psihiatrie, Socola, Iași, Iaşi
  - Jebel, Timuș, Jebel Timis
  - Spitalul Clinic de Psihiatrie, "Ghe. Preda" Sibiu, Sibiu, Sibiu County
  - Spitalul Clinic de Urgenta Clinica "E. Pamfil", Timișoara, Timisoara
  - Spitalul Clinic de Psihiatrie, sectia 14, Berceni St., 10-12, Bucharest
  - Spitalul Clinic de Psihiatrie, sectia 10, Berceni St., 10-12, Sector 4, Bucharest
  - Spitalul Clinic, sectia 8, Berceni St., Sector 4 Bucharest
  - Spitalul de Psihiatrie, Titan, Bld Nicolae Grigorescu, No. 41, Sector 3,
  - Spitalul Clinic de Psihiatrie "Prof.Al. Obregia" Sectia 11, Bucharest
  - Spitalul Clinic Judetean De Urgenta, Clinica Psihiatrie, Octavian Goga St, 17, Arad
  - Spitalul de Psihiatrie Botosani, Str. I.C.Bratianu Nr. 116, Botosani
  - Spitalul Clinic Judetean, Sectia Clinica Psihiatrie, Str. Victor Babes, Nr. 43, Cluj Napoca
  - Spitalul de Psihiatrie si Neurologie, Str.Mihai Eminescu, Nr.18, Brasov